CLINICAL TRIAL: NCT02747498
Title: Comparison of Circumferential Pulmonary Vein Isolation and Complex Pulmonary Vein Isolation Additional Linear Ablation for Recurred Atrial Fibrillation After Previous Catheter Ablation: Prospective Randomized Trial
Brief Title: Comparison of Circumferential Pulmonary Vein Isolation and Complex Pulmonary Vein Isolation Additional Linear Ablation for Recurred Atrial Fibrillation After Previous Catheter Ablation: Prospective Randomized Trial (RILI Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-1057
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Recurred Atrial Fibrillation
Keywords: Recurred atrial fibullation; CPVI; posterior wall isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- circumferential pulmonary vein isolation (Active Comparator): Procedure with circumferential pulmonary vein isolation for atrial fibrillation
  Interventions: Procedure: Procedure with circumferential pulmonary vein isolation
- Posterior box isolation in addiction to pulmonary vein isolation (Experimental): Posterior box isolation in addiction to circumferential pulmonary vein isolation
  Interventions: Procedure: Procedure with linear ablation in addiction to pulmonary vein isolation

INTERVENTIONS:
Procedure: Procedure with circumferential pulmonary vein isolation — We will compare circumferential pulmonary vein (PV) isolation (CPVI) alone and posterior box isolation in addition to CPVI in patients with AF recurrence after de novo ablation procedures and with PV reconnections with 1:1 randomization. We will conduct ablation procedures by 3D electroanatomical mapping guidance and confirm bidirectional blocks of each ablation lines by differential pacing. For posterior box isolation, we will ablate remaining atrial potentials with point by point ablation to avoid the risk of esophageal injury at posterior inferior line. In all patients, mapping and ablation for non-pulmonary vein foci will be done with isoproterenol infusion at the end of the procedure. We will compare procedure time, ablation time, procedure related complication rates, and clinical recurrence rate of AF during follow-up period.
  Arms: circumferential pulmonary vein isolation
Procedure: Procedure with linear ablation in addiction to pulmonary vein isolation — We will compare circumferential pulmonary vein (PV) isolation (CPVI) alone and posterior box isolation in addition to CPVI in patients with AF recurrence after de novo ablation procedures and with PV reconnections with 1:1 randomization. We will conduct ablation procedures by 3D electroanatomical mapping guidance and confirm bidirectional blocks of each ablation lines by differential pacing. For posterior box isolation, we will ablate remaining atrial potentials with point by point ablation to avoid the risk of esophageal injury at posterior inferior line. In all patients, mapping and ablation for non-pulmonary vein foci will be done with isoproterenol infusion at the end of the procedure. We will compare procedure time, ablation time, procedure related complication rates, and clinical recurrence rate of AF during follow-up period.
  Arms: Posterior box isolation in addiction to pulmonary vein isolation

SUMMARY:
The purpose of this study is to compare the clinical outcomes depending on catheter ablation strategy for repeat ablation procedure among the patients with recurred atrial fibrillation after de novo catheter ablation. After randomization, we will conduct circumferential pulmonary vein isolation alone in a group, and additional posterior box isolation in the other group. Non-pulmonary vein foci ablation will be done in all patients. We will compare clinical recurrence rate, complication rate, and procedure time, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AF aged between 20 and 80 years old.
2. Patients possible to anticoagulation and anti arrhythmic drug
3. Patients who had undergone de novo ablation procedures based on circumferential pulmonary vein isolation with no additional linear ablations
4. Patients undergoing a second ablation procedure due to clinical recurrence resistant to antiarrhythmic drugs with findings of PV reconnections

Exclusion Criteria:

1. Structural cardiac disease 2. Contraindication to brain perfusion CT 3. Catheter ablation history for AF, Cardiac surgery for AF 4. active internal bleeding 5. Impossible to anticoagulation or antiarrhythmic drug 6. valvular AF ((MA> GII, Mechanical valve, Mitral valve raplacement) 7. Patients with severe medical disease 8. Expected survival < 1year 9. Severe alcoholics, drug addiction 10. Pregnancy 11. LA diameter>60mm

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Clinical recurrence of atrial fibrillation after catheter ablation | 3 years
  We defined recurrence of AF as any episode of AF or atrial tachycardia lasting longer than 30 sec. Any ECG documentation of AF recurrence after 3 months was diagnosed as clinical recurrence.

SECONDARY OUTCOMES:
procedure time | 1 day
procedure related complication rate | 3 years
rate of hospitalization | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SJ, Yu HT, Choi SH, Kim D, Kim TH, Uhm JS, Joung B, Lee MH, Pak HN. Extended Period Outcomes of Posterior Box Isolation in 4 Randomized Atrial Fibrillation Catheter Ablation Trials. JACC Asia. 2025 Feb;5(2):285-295. doi: 10.1016/j.jacasi.2024.12.002. Epub 2025 Feb 4. PMID 39967220
- [Derived] Kim D, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Pak HN. Electrical Posterior Box Isolation in Repeat Ablation for Atrial Fibrillation: A Prospective Randomized Clinical Study. JACC Clin Electrophysiol. 2022 May;8(5):582-592. doi: 10.1016/j.jacep.2022.01.003. Epub 2022 Feb 23. PMID 35589170